CLINICAL TRIAL: NCT05172934
Title: Adjunctive Intra-arterial Tenecteplase Following Mechanical Thrombectomy Pilot Trial
Acronym: ALLY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ProMedica Health System (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALLY
Record Dates: First submitted 2021-11-16; First posted 2021-12-29 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Ischemic Stroke
Keywords: thrombolytic; stroke; distal emboli
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Intervention Model Description: Participants will receive intra-arterial Tenecteplase after achieving mTICI 2b or 2c reperfusion with standard of care mechanical thrombectomy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intra-arterial Tenecteplase (Experimental): Participants will receive intra-arterial Tenecteplase after achieving mTICI 2b or 2c reperfusion with standard of care MT.
  Interventions: Drug: intra-arterial tenecteplase

INTERVENTIONS:
Drug: intra-arterial tenecteplase — intra-arterial drug administered after mechanical thrombectomy

SUMMARY:
Prospective, single center, non-randomized, pilot study to assess the feasibility of IA TNK following standard of care mechanical thrombectomy (MT) in patients with AIS. Participants will receive IA TNK after achieving mTICI 2b or 2c reperfusion with standard of care MT. Patients enrolled into the study will be followed for 3 months after treatment with IA TNK.

DETAILED DESCRIPTION:
As current MT technology is not amenable to retrieval of distal occlusions (M3/M4, etc), we hypothesize that IA lytic may play an important role as an adjunctive therapy to open up distal vessels (after the primary LVO has been removed) to achieve complete or near complete reperfusion. In this pilot trial, our goal is to assess the feasibility and safety of IA Tenecteplase (TNK) as an adjunctive therapy following standard of care mechanical thrombectomy (MT) in patients with AIS. A total of 20 patients will be enrolled into the ALLY pilot study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-85
* 2. Anterior circulation ischemic stroke symptoms with confirmed occlusion (ICA, M1, or M2) on angiogram and mechanical thrombectomy initiated within 24 hours since last known well
* 3. a. Patients treated less than 6 hours since last known well with ASPECTS >6. b. Patients treated beyond 6 hours since last known well, CT or MRI perfusion scan showing favorable mismatch profile (Target mismatch profile on CT perfusion or MRI (ischemic core volume is <70ml, mismatch ratio is >1.8 and mismatch volume is >15ml)
* 4. Post-mechanical thrombectomy with ≤5 device passes and mTICI grade 2b or 2c with persistent occlusion(s) in terminal branches not amenable to MT.
* 5. Signed informed consent

Exclusion Criteria:

* 1. Premorbid modified Rankin scale (mRS) score of 4 or greater
* 2. Presence of any hemorrhage and/or ASPECT score ≤6 on baseline head CT
* 3. Platelet count <100,000
* 4. Known bleeding diathesis
* 5. Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency
* 6. Active anticoagulation treatment with novel oral anticoagulant (NOACs) taken within the last 48 hours, or INR >1.8
* 7. Patients requiring active treatment with dual antiplatelet agents (e.g. proximal cervical carotid artery stenting)
* 8. Pregnant or lactating
* 9. Previous known allergy to TNK
* 10. Major surgery in past 30 days
* 11. Patient is on or requires dialysis
* 12. History of intracranial hemorrhage or serious head trauma at any time
* 13. Any condition in the opinion of the enrolling physician that would preclude the patient from participating
* 14. Pre-existing medical, neurological, or psychiatric disease that would confound the neurological or functional evaluation
* 15. Severe, uncontrolled hypertension (systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg) that is refractory to treatment
* 16. History of acute ischemic stroke in the last 60 days
* 17. Presumed septic embolus; suspicion of bacterial endocarditis
* 18. Suspicion of aortic dissection
* 19. Intracranial neoplasm
* 20. Any mass effect
* 21. Any terminal medical condition with life expectancy less than 6 months
* 22. Concurrent enrollment in another trial that could confound the results of this study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Incidence of any intracranial hemorrhage and neurologic worsening | 24 hours post-treatment with intra-arterial Tenecteplase
  Incidence of any intracranial hemorrhage and neurologic worsening of at least 4 points on the National Institute of Health Stroke Scale (NIHSS), according to the European Cooperative Acute Stroke Study II (ECASS-II) criteria, within 24 hours of treatment with IA TNK

SECONDARY OUTCOMES:
Improved reperfusion | immediate post-treatment
  Proportion of patients with improved reperfusion (mTICI 2c/3) at end of IA treatment
Improved reperfusion | immediate post-treatment
  Proportion of patients with improvement of reperfusion to mTICI 2c, mTICI 3, and mTICI 2c-3.
Ordinal modified Rankin Scale Score | 90 days post-treatment
  Ordinal modified Rankin Scale Score at 90 days. The mRS is the standard tool to assess neurological outcome in trials with acute severe brain disease. The scale runs from 0-6, running from perfect health without symptoms (= 0) to death (= 6).
Functional Independence | 90 days post-treatment
  Proportion of patients with functional independence, defined as a mRS of 0-2 at 90 days
Final revascularization grade | immediate post-treatment
  Final revascularization grade at end of IA treatment using the modified Thrombolysis in Cerebral Infarction (mTICI) grading scale.
Mortality | Hospital Discharge (Day 6 post-randomization (+/- 1 day))
  Mortality rate at discharge
Asymptomatic intracranial hemorrhage | 24 hours post-treatment
  Incidence of any asymptomatic intracranial hemorrhage
Mean number of boluses | Immediate post-procedure
  Mean number of boluses to achieve improvement in reperfusion to mTICI 2c and mTICI 3

CONTACTS AND LOCATIONS:
Overall Officials: Syed F Zaidi, MD, Principal Investigator — ProMedica Health System
Locations (1):
- ProMedica Toledo Hospital, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zaidi SF, Castonguay AC, Zaidat OO, Jadhav AP, Sheth SA, Haussen DC, Nguyen TN, Burgess RE, Alhajala HS, Gharaibeh K, Salahuddin H, Rao R, Oliver MJ, Jumaa MA. Safety of Adjunctive Intraarterial Tenecteplase Following Mechanical Thrombectomy: The ALLY Pilot Trial. Stroke. 2025 Feb;56(2):355-361. doi: 10.1161/STROKEAHA.124.048846. Epub 2025 Jan 8. PMID 39772606